CLINICAL TRIAL: NCT06235372
Title: Evaluation of the Corneal Endothelial Cell Layer by Specular Microscopy in Patients With Thyroid Eye Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mayar Ashraf Mohamed, Principal investigator, Assiut University
Other Study IDs: Specular microscopy in TED
Record Dates: First submitted 2023-12-22; First posted 2024-01-31 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-01

CONDITIONS: Thyroid Eye Disease
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Specular microscopy — Specular microscopy is a noninvasive photographic technique that analyze the corneal endothelium. Using computer-assisted morphometry, modern specular microscopes analyze the size, shape and population of the endothelial cells. The instrument projects light onto the cornea and captures the image that is reflected from the optical interface between the corneal endothelium and the aqueous humor. The reflected image is analyzed by the instrument and displayed as a specular photomicrograph .

SUMMARY:
To investigate corneal endothelial cell layer damage by specular microscopy in patients with thyroid eye disease

DETAILED DESCRIPTION:
Thyroid eye disease is a common periorbital autoimmune inflammatory disease .It significantly impairs quality of the life ,causes cosmetic defects ,and could be sight-threatening ,especially when optic nerve or the cornea is affected.Classic manifestations of thyroid eye disease include proptosis ,lid retraction ,lagophthalmos,optic neuropathy and restrictive extraocular myopathy.In addition to the affection of the orbital and lacrimal glands ,the corneal endothelium has showen morphological changes in patients with thyroid eye disease .corneal endothelium is the innermost corneal layer facing the anterior chamber and is known for maintaining corneal transparency by its pump-leak function .corneal transparency is crucial for optimal vision . severe damage to corneal endothelium can induce corneal opacification .resulting in corneal edema and subsequently vision loss. That is because there are thyroxine receptors in all layers of the conea. And the autoantibodies to TSH receptors usually attach to them causing damage to the cornea.Specular microscopy is one of the best investigative procedure used to assess changes in the corneal endothelium due to thyroid eye disease.Specular microscopy is a noninvasive photographic technique that analyze the corneal endothelium. Using computer-assisted morphometry, modern specular microscopes analyze the characteristics of the endothelial cells. The instrument projects light onto the cornea and captures the image that is reflected from the optical interface between the corneal endothelium and the aqueous humor. The reflected image is analyzed by the instrument and displayed as a specular photomicrograph

ELIGIBILITY:
Inclusion Criteria:

* Patients with thyroid eye disease whom diagnosis was established based on bartley diagnostic criteria .

Exclusion Criteria:

* participates with systemic diseases other than HT such as

  1. diabetes mellitus
  2. previous ocular surgery or laser therapy.
  3. history of corneal disease.
  4. history of trauma.
  5. history of glaucoma

Ages: 12 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with thyroid eye disease whom diagnosis was established based on bartley diagnostic criteria .
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-03-21 (Estimated); Primary Completion 2025-10-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Damage of the corneal endothelial cells in patients with thyroid eye disease by specular microscopy | Baseline
  To detect if there is any change in corneal endothelial cell layer in patients with thyroid eye disease

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Mohammed, Professor, Study Director — Academic organizations; Khaled Abdelazim, Assistant professor, Study Director — Academic organizations; Ahmed Abdelnasser, Lecturer, Study Director — Academic organizations